CLINICAL TRIAL: NCT03706196
Title: Comparison of Environmental Factors Between the Areas of Over- and Under-incidence of Crohn's Disease in the Haut de France Region, by the Study of Dental Exposomes
Acronym: EXPOSOMES
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_44; 2018-A00195-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Environmental Exposure
Keywords: dental exposome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high incidence crohn's disease area: subjects living in high incidence crohn's disease area coming in dentist for dental extraction linked to medical indication
- low incidence crohn's disease area: subjects living in low incidence crohn's disease area coming in dentist for dental extractionlinked to medical indication

SUMMARY:
the aim of this preliminary observational study is to compare external exposomes from 10 teeth issued through 10 subjects living in high incidence of crohn's disease area and 10 teeth issued through 10 subjects living in low incidence of crohn's disease area.

ELIGIBILITY:
Inclusion Criteria:

* adults subjects living in high and low incidence of crohn's disease areas and needing a dental extraction for medical indication

Exclusion Criteria:

* smokers during 10 last years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults subjects living in high and low incidence of crohn's disease areas and needing a dental extraction for medical indication.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
comparison of aluminum rate using metabolomic method in teeth between subjects living in high and low incidence crohn's disease areas. | Baseline: one session

SECONDARY OUTCOMES:
comparison of environmental exposomes using metabolomic method in teeth between subjects living in high and low incidence crohn's disease areas. | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: Corinne GOWER, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France